CLINICAL TRIAL: NCT04448639
Title: STAMI- Stunning in Takotsubo Versus Acute Myocardial Infarction
Brief Title: Stunning in Takotsubo Versus Acute Myocardial Infarction
Acronym: STAMI
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Björn Redfors, Doctor of medicine, PhD; Associate Proffessor, Vastra Gotaland Region
Other Study IDs: Dnr 2019-04092
Record Dates: First submitted 2020-06-03; First posted 2020-06-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Myocardial Stunning
Keywords: Myocardial Stunning; Acute heart failure; Taoktsubo Syndrome; Acute myocardial infarction
MeSH Terms: conditions — Myocardial Stunning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STEMI: Patients with ST-elevation myocardial Infarction (STEMI) (TS) who undergo urgent coronary angiography within 12 hours of symptom onset.
  Interventions: Diagnostic Test: Echocardigraphy (ECHO); Diagnostic Test: Bloodtest
- TS: Patients with Takotsubo Syndrome (TS) who undergo urgent coronary angiography within 12 hours ofsymptom onset.
  Interventions: Diagnostic Test: Echocardigraphy (ECHO); Diagnostic Test: Bloodtest

INTERVENTIONS:
Diagnostic Test: Echocardigraphy (ECHO) — Standar 12 lead electrocardiogram
  Other Names: Standard electrocardigraphy (ECG )
Diagnostic Test: Bloodtest — cardiac biomarkers
  Other Names: Troponin and NT-proBNP

SUMMARY:
The Stunning in Takotsubo versus Acute Myocardial Infarction (STAMI) Study

Background: Acute myocardial stunning, herein defined as the reversible loss of myocardial function, occurs in both takotsubo syndrome (TS) and ST-elevation myocardial infarction (STEMI), and can be life-threatening in both conditions. However, despite typically having considerably more pronounced myocardial stunning, TS patients have better prognosis than patients with STEMI. Despite the different relationship between extent of myocardial stunning and prognosis in TS vs STEMI, no 'head-to-head' comparison of the myocardial stunning phenotypes in TS vs STEMI has been done.

Methods: The Stunning In Takotsubo and Acute Myocardial Infarction (STAMI) study is a single-center, prospective clinical study that will enroll 100 patients with STEMI and 25 patients with TS. Echocardiography, laboratory testing (including troponin and NTpro-BNP), and ECG will be done immediately after angiography and at days 1, 2, 3, 7, 14 and 30. The primary endpoint is the proportion of myocardial stunning that has resolved after 72 hours, as determined by echocardiography. Total myocardial stunning is defined as the extent of akinesia observed at day 0 that resolves by day 30.

DETAILED DESCRIPTION:
Prospective assessment of the temporal electrocardiographic-, vectorcardiographic- and echocardiographic changes in STelevation myocardial infarction versus the takotsubo syndrome.

AIM To compare the temporal pattern of myocardial funtional recovery after ST-elevation myocardial infarction (STEMI) versus the takotsubo syndrome (TS).

BACKGROUND Modern therapies have reduced the incidence of acute ischemic heart failure (AIHF) -But AIHF is still common and once it develops prognosis remains dismal.Despite considerable therapeutic advancements over the last decades, acute myocardialinfarction (AMI) remains one of the most common causes of death . Among patients who are admitted with AMI, the 10% that develop AIHF account for approximately 50% of Deaths within 30 days . The prognosis for patients with AIHF has not improved over the last decade . AIHF occurs due to acute loss of cardiac function, some of which occurs in myocardium that is not irreparably damaged - so called stunned myocardium.

Myocardial stunning in AIHF - Temporary mechanical dysfunction without irreparable injury. Myocardial stunning was originally described in the setting of ischemia and was defined as temporary mechanical dysfunction that persists after resolution of ischemia, with the absence of irreversible histological damage . For the purpose of this application it is more broadly defined as temporary mechanical dysfunction, with the absence of irreversible histological damage - irrespective of the underlying cause. Myocardial stunning is believed to be a harmful phenomenon caused by cellular injury .

Study hypothesis: Myocardial stunning is a protective mechanism by which the cardiomyocytes preserve energy for vital processes in states of severe cellular stress - but that can "overshoot" and lead to potentially lethal cardiac decompensation. In the normal heart, the contractile apparatus consumes the majority of myocardial energy and oxygen . Non-contractile myocardial functions, including cellular and electrical homeostasis, require less than 20% as much oxygen. When oxygen supply to the heart is interrupted myocardial stunning ensues within seconds, whereas it takes at least 10 minutes for the cardiomyocyte's energy metabolites to decrease to 50% of their initial level .Hence, by shutting down the contractile apparatus before it consumes the cells' energy stores myocardial stunning effectively preserves energy for processes that are necessary for cell survival . Irrespective of its beneficial effects on cardiomyocyte metabolism, myocardial stunning may lead to sufficiently pronounced cardiac dysfunction to cause life-threatening AIHF.

Study purpose:

To better understand the difference between myocardial stunning in STEMI and the more benign form of stunning in TS. The sudden occurrence of temporary myocardial mechanical dysfunction with the absence of irreversible myocardial damage is not limited to AMI. It can occur postoperatively after cardiac arrest; in the settings of acute myocarditis and tachycardia-induced cardiomyopathy; and as a consequence of severe emotional or somatic stress in the takotsubo syndrome .Intriguingly, takotsubo is characterized by a compensated hemodynamic profile despite extensive myocardial dysfunction, effective recovery of myocardial function within days orweeks, and a relatively good prognosis .Takotsubo therefore appears to be a more efficient form of stunning than AIHF. Better understanding of the mechanisms behind the stunning phenomenon could allow for manipulation of the stunning phenotype in AIHF, or for pharmacological reversal of myocardial stunning once coronary reperfusion and adequate myocardial energy delivery has been ensured.

ELIGIBILITY:
Inclusion Criteria:

* STEMI or TS with planned coronary angiography within 12 hours from the onset of symptoms
* Written consent

Exclusion Criteria:

* Cardiogenic shock, defined as Killip class IV
* Expected inability to comply with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with STEMI or TS who undergo urgent coronary angiography within 12 hours of symptom onset.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of stunning that has resolved at 3 days versus 14 days | 30 days
  StunningResolution at 3 days is defined as StunningRes3D = (%Akinesia Baseline - %Akinesia 3day) / (%Akinesia Baseline -
  %Akinesia 30days); where %Akinesia is calculated as the endocardial length of the akinetic left ventricular myocardium divided by the total endocardial length of the left ventricular myoocardium - as assessed in the apical 2-chamber and 4-chamber views at end-diastole.
  The recovery of stunning at 3 days is compared to the recovery of stunning at 30 days. Thus a 14 day timeframe is required.

SECONDARY OUTCOMES:
Change in wall motion score index | 30 days
  Myocardial wall motion score index
Change in left ventricular ejection fraction | 30 days
  left ventricular ejection fraction as measured by speckle tracking echocardiography.
Change in global longitudinal strain | 30 days
  Global longitudinal strain as measured by speckle tracking echocardiography.
Change in radial strain in the unaffected contralateral myocardial wall | 30 days
  Radial longitudinal strain as measured by speckle tracking echocardiography.
Change in serum troponin-I:troponin:T ratio | 30 days
  The ratio between serum troponin-1 and serum troponin-T
Change in serum NT proBNP | 30 days
  Serum NT proBNP

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology; Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jha S, Poller A, Shekka Espinosa A, Molander L, Sevastianova V, Zeijlon R, Simons K, Bobbio E, Pirazzi C, Martinsson A, Mellberg T, Gudmundsson T, Torild P, Sundstrom J, Andersson EA, Thorleifsson S, Salahuddin S, Elmahdy A, Pylova T, Rawshani A, Angeras O, Ramunddal T, Skoglund K, Omerovic E, Redfors B. Prospective comparison of temporal changes in myocardial function in women with Takotsubo versus anterior STEMI. Clin Res Cardiol. 2025 Dec;114(12):1705-1717. doi: 10.1007/s00392-025-02633-4. Epub 2025 Mar 20. PMID 40111441